CLINICAL TRIAL: NCT04978363
Title: Effects of a Hands Free Crutch on Walking Stability During Gait
Brief Title: iWalk Hands Free Crutch
Acronym: HFC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Collaborators: iWalkFree, Inc. (Industry)
Responsible Party: Principal Investigator, Jason Wilken, Associate Professor of Physical Therapy and Rehabilitation Science, University of Iowa
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 202101408
Record Dates: First submitted 2021-07-18; First posted 2021-07-27 (Actual); Results first posted 2023-05-22 (Actual); Last update posted 2023-05-22 (Actual); Status verified 2023-04

CONDITIONS: Healthy
Keywords: Hands Free Crutch; Crutches; Assistive devices; Balance; Walking stability; Gait analysis; Adult; Biomechanics; Walking boot
MeSH Terms: interventions — Crutches

STUDY DESIGN:
Intervention Model Description: All participants will complete all six testing conditions, including:
  1. BOOT (walking boot)
  2. HFC + BOOT (Hands Free Crutch with the walking boot)
  3. SAC + BOOT (Standard Axillary Crutches with the walking boot)
  4. NONE (no device/baseline)
  5. HFC NO BOOT (Hands Free Crutch with no walking boot) and
  6. SAC NO BOOT (Standard Axillary Crutches with no walking boot).
  The order of the four primary conditions will be randomized using an online random number generator (1-4) with:
  1=NONE, 2=BOOT only, 3=HFC+BOOT, and 4=SAC+BOOT.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (6):
- Arm 1. NONE (No Intervention): Participants will be tested while wearing no boot and no assistive device.
- Arm 2. BOOT (Experimental): The first intervention condition tested is a walking boot only on the subject's right lower extremity.
  Interventions: Device: BOOT
- Arm 3. HFC+BOOT (Experimental): The second intervention condition tested is a Hands Free Crutch (HFC) with the walking boot, both worn on the subject's right lower extremity.
  Interventions: Device: HFC+BOOT
- Arm 4. SAC+BOOT (Experimental): The third intervention condition tested is standard axillary crutches (SAC) with the walking boot worn in non-weight bearing on the subject's right lower extremity.
  Interventions: Device: SAC+BOOT
- Arm 5. HFC (Experimental): The fourth intervention condition tested is the Hands Free Crutch worn on the subject's right lower extremity without the walking boot.
  Interventions: Device: HFC
- Arm 6. SAC (Experimental): The fifth and last intervention condition tested is standard axillary crutches with the subject non-weight bearing on the right lower extremity without the walking boot.
  Interventions: Device: SAC

INTERVENTIONS:
Device: BOOT — A walking boot is a common type of brace/boot that restricts ankle and foot movement.
  Other Names: Walking Boot; CAM Boot; Controlled Ankle Motion Boot
  Arms: Arm 2. BOOT
Device: HFC — The Hands Free Crutch (HFC) by iWalkFree, Inc. is a novel, ambulatory assistive device that prevents foot and ankle loading while also allowing free use of the arms and hands.
  Other Names: Hands Free Crutch; iWalk Free; iWalk 3.0
  Arms: Arm 5. HFC
Device: SAC — Standard axillary crutches (SAC) are ambulatory assistive devices, commonly used for lower extremity injuries or surgeries.
  Other Names: Standard Axillary Crutches; axillary crutches; crutches; underarm crutches
  Arms: Arm 6. SAC
Device: HFC+BOOT — The Hands Free Crutch (HFC) by iWalkFree, Inc. is a novel, ambulatory assistive device that prevents foot and ankle loading while also allowing free use of the arms and hands. A walking boot is a common type of brace/boot that restricts ankle and foot movement.
  Arms: Arm 3. HFC+BOOT
Device: SAC+BOOT — Standard axillary crutches (SAC) are ambulatory assistive devices, commonly used for lower extremity injuries or surgeries. A walking boot is a common type of brace/boot that restricts ankle and foot movement.
  Arms: Arm 4. SAC+BOOT

SUMMARY:
The proposed study evaluates the effects of a hands free crutch (iWalkFree, Inc.) on walking balance and stability compared to standard crutches. It is expected that the hands free crutch will provide better stability during walking on a level surface and better reported balance confidence compared to standard crutches. In this study, walking stability will be assessed using motion capture data from an infrared camera system with 12 mounted cameras surrounding a level walkway. Balance will be assessed through a self-reported activity-specific balance confidence (ABC) questionnaire. An improved understanding of the effects of the hands free crutch on gait may benefit the future prescription of ambulatory assistive devices. The proposed study may provide insight that can be used by physical therapists and other providers to select the ambulatory assistive device that best meets their patients' needs.

DETAILED DESCRIPTION:
The purpose of this study is to compare the hands free crutch (HFC) to standard axillary crutches (SACs) with and without a walking boot, using outcomes related to walking stability, balance confidence, patient preference, device comfort, and any reported pain while using the devices.

Healthy, able-bodied individuals will wear a walking boot to simulate a below knee injury or post-surgery condition during participation. They will maintain a non-weight bearing status while completing the 4 research conditions in randomized order: 1) BOOT, 2) HFC + BOOT, 3) SAC + BOOT, or 4) NONE.

Participants will complete 5 total sessions, with 4 biomechanics data collection sessions corresponding to the 4 conditions. At the first visit, participants will complete pre-consent screening and consent paperwork. Then they will be randomized to the 4 conditions above, and anthropometric (body height, weight/mass, leg length, shoe length and width) and demographic data will be collected. Participants will accommodate overnight to each of the 4 study conditions before testing. If participants are randomized to the NONE condition first, they will have the option of completing testing in that condition (no Boot) at the initial visit. The primary dependent measure is whole body angular momentum, an objective measure of walking stability.

Data will be collected using over 50 small reflective markers placed on the participants and the assistive devices, a computerized motion capture system and force plates embedded in the floor. The force plates capture ground reaction forces which will be used to calculate joint moments for interpretation of angular momentum data. The motion capture system will be used to evaluate joint and segment kinematics and temporal-spatial data to characterize the gait pattern in each condition and calculate angular momentum.

The second purpose of this research study is to determine the effect of crutch use on participant reported balance confidence and device preference. A validated balance confidence questionnaire and participant satisfaction, comfort and preference will be used to compare between conditions. A numerical pain rating scale (0-10) will be used to assess for any reported pain in all of the conditions.

The third purpose of this research is to determine the effect of crutch (HFC and SACs) and boot (with and without) use on walking stability as measured by whole body and segmental angular momentum during gait. Two additional conditions are added to address this purpose (HFC NO BOOT and SAC NO BOOT), resulting in a total of 6 research conditions:

1) BOOT, 2) HFC + BOOT, 3) SAC + BOOT 4) NONE, 5) HFC NO BOOT, 6) SAC NO BOOT The HFC NO BOOT condition will be evaluated at the end of the HFC + BOOT session, and the SAC NO BOOT condition will be evaluated at the end of the SAC + BOOT session to stay within the fiscal and logistical constraints of the project. Previously described methods will be used.

Ultimately, this study could assist physical therapists and other providers in the clinical prescription and application of such devices.

ELIGIBILITY:
Inclusion Criteria:

* Male or Female
* Ages: 18 - 45
* Height between 5'2" and 6'6"
* Foot size that corresponds to available walking boots
* Healthy individuals without current complaint of lower extremity pain, spine pain, open wounds or active infection
* Full active pain free range of motion of the bilateral upper and lower extremities and spine
* Able to hop without pain
* Able to perform a full squat without pain
* Able to walk up and down a flight of stairs at normal walking speed without using the hand rail
* Able to stand on one leg for at least 30 seconds
* Able to read and write in English and provide written informed consent

Exclusion Criteria:

* Weight greater than 270 lbs
* BMI greater than 35
* Maximum thigh circumference at top of the leg greater than 28"
* Prior medical or neuromusculoskeletal disorders that have limited their participation in work or exercise in the last 6 months
* Prior lower extremity injury proximal to the ankle requiring surgery or limiting function for greater than 6 weeks
* Prior back pain that recurs or has limited activities for greater than 6 weeks
* Diagnosed moderate or severe brain injury
* Diagnosis of a physical or psychological condition that would preclude testing (e.g. cardiac condition, clotting disorder, pulmonary condition)
* Uncorrected visual or hearing impairment(s)
* Require use of an assistive device
* Pregnancy - Per participant self-report. Due to the expected small number of pregnant individuals, and resulting inability to account for its effect on resulting outcomes, participants will be withdrawn from the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2021-10-05 (Actual); Primary Completion 2022-01-27 (Actual); Study Completion 2022-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jason M Wilken, PT, PhD, Principal Investigator — University of Iowa, Department of Physical Therapy and Rehabilitation Science
Locations (1):
- Human Performance and Clinical Outcomes Lab, The University of Iowa, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited by mass email and postings on a university news website between September 2021 and January 2022. The first participant was enrolled on October 5, 2021, and the last participant was enrolled on January 16, 2022.
Pre-assignment Details: One participant was enrolled in the study and then failed the post-screening. As a result they were excluded before assignment to the groups.
Groups:
- NONE, HFC+BOOT, SAC+BOOT, BOOT; NONE, BOOT, SAC+BOOT, HFC+BOOT; NONE, SAC+BOOT, BOOT, HFC+BOOT; NONE, BOOT, HFC+BOOT, SAC+BOOT; SAC+BOOT, NONE, BOOT, HFC+BOOT; SAC+BOOT, BOOT, NONE, HFC+BOOT; BOOT, NONE, SAC+BOOT, HFC+BOOT; BOOT, NONE, HFC+BOOT, SAC+BOOT; BOOT, HFC+BOOT, NONE, SAC+BOOT; HFC+BOOT, BOOT, NONE, SAC+BOOT; HFC+BOOT, NONE, BOOT, SAC+BOOT: The testing order of each of four primary conditions (BOOT, HFC + BOOT, SAC + BOOT, or NONE) will be randomized for each participant.
Period: Overall Study
Arm/Group | NONE, HFC+BOOT, SAC+BOOT, BOOT | NONE, BOOT, SAC+BOOT, HFC+BOOT | NONE, SAC+BOOT, BOOT, HFC+BOOT | NONE, BOOT, HFC+BOOT, SAC+BOOT | SAC+BOOT, NONE, BOOT, HFC+BOOT | SAC+BOOT, BOOT, NONE, HFC+BOOT | BOOT, NONE, SAC+BOOT, HFC+BOOT | BOOT, NONE, HFC+BOOT, SAC+BOOT | BOOT, HFC+BOOT, NONE, SAC+BOOT | HFC+BOOT, BOOT, NONE, SAC+BOOT | HFC+BOOT, NONE, BOOT, SAC+BOOT
Started | 2 | 2 | 2 | 1 | 3 | 1 | 2 | 2 | 2 | 2 | 1
Discontinued Intervention | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 2 | 1 | 1 | 1 | 2 | 1 | 2 | 2 | 2 | 2 | 1
Not Completed | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other medical issues unrelated to the study | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Unable to meet the necessary time commitment | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Didn't feel safe and had pain with hands-free crutch | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NONE, HFC+BOOT, SAC+BOOT, BOOT | NONE, BOOT, SAC+BOOT, HFC+BOOT | NONE, SAC+BOOT, BOOT, HFC+BOOT | NONE, BOOT, HFC+BOOT, SAC+BOOT | SAC+BOOT, NONE, BOOT, HFC+BOOT | SAC+BOOT, BOOT, NONE, HFC+BOOT | BOOT, NONE, SAC+BOOT, HFC+BOOT | BOOT, NONE, HFC+BOOT, SAC+BOOT | BOOT, HFC+BOOT, NONE, SAC+BOOT | HFC+BOOT, BOOT, NONE, SAC+BOOT | HFC+BOOT, NONE, BOOT, SAC+BOOT | Total
Number analyzed (Participants) | 2 | 2 | 2 | 1 | 3 | 1 | 2 | 2 | 2 | 2 | 1 | 20
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 2 | 1 | 3 | 1 | 2 | 2 | 2 | 2 | 1 | 20
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 27 (7.8) | 19 (1.4) | 27 (12.0) | 41 (0.0) | 27 (6.7) | 27 (0.0) | 32 (14.1) | 23 (3.5) | 21 (3.5) | 32 (1.4) | 18 (0.0) | 27 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 1 | 0 | 2 | 1 | 1 | 2 | 1 | 0 | 1 | 12
  Male | 0 | 1 | 1 | 1 | 1 | 0 | 1 | 0 | 1 | 2 | 0 | 8
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 2 | 2 | 1 | 3 | 1 | 2 | 1 | 1 | 2 | 1 | 18
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 2 | 2 | 1 | 1 | 3 | 1 | 2 | 1 | 1 | 1 | 1 | 16
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Whole Body Angular Momentum-sagittal Plane
Description: Range of whole-body angular momentum in the sagittal plane during gait using the motion capture system. While angular momentum can be measured in kg*m^2/second it is reported as dimensionless in this study as it has been normalized to body weight (kg), height (m), and walking speed (m/s).
Time Frame: one session (up to 2 hours long), out of 4 total sessions
Population: Healthy able-bodied individuals
Measure: Mean (Standard Deviation); unit: dimensionless
Arm/Group | Arm 1. NONE | Arm 2. BOOT | Arm 3. HFC+BOOT | Arm 4. SAC+BOOT | Arm 5. HFC | Arm 6. SAC
Number analyzed (Participants) | 17 | 17 | 17 | 17 | 17 | 17
dimensionless | 0.051 (0.009) | 0.079 (0.011) | 0.095 (0.010) | 0.155 (0.033) | 0.077 (0.011) | 0.142 (0.027)

2. Other Pre Specified Outcome: Activity-specific Balance Confidence (ABC) Scale
Description: Balance confidence will be assessed using the ABC Scale on 16 activities, using a 0-100% scale (0% = no confidence and 100% = completely confident).
Time Frame: Baseline
Population: Healthy able-bodied individuals completed the outcome measure for the arms listed above. They did not complete the outcome measure for HFC+Boot and SAC+Boot.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Arm 1. NONE | Arm 2. BOOT | Arm 5. HFC | Arm 6. SAC
Number analyzed (Participants) | 17 | 17 | 17 | 17
score on a scale | 98.75 [95.94 to 100.00] | 87.50 [77.50 to 93.13] | 57.50 [45.94 to 70.31] | 58.82 [44.69 to 72.81]

3. Other Pre Specified Outcome: Numerical Pain Rating Scale
Description: Pain will be assessed using a standard 11-point numerical pain rating scale, in which 0 = no pain and 10 = worst pain imaginable.
Time Frame: over three sessions (an average of 2 hours for each session)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Arm 1. NONE | Arm 2. BOOT | Arm 5. HFC | Arm 6. SAC
Number analyzed (Participants) | 17 | 17 | 17 | 17
units on a scale | 0.00 (0.00) | 1.12 (1.76) | 2.59 (1.73) | 2.47 (1.91)

4. Other Pre Specified Outcome: Participant Device Comfort Score
Description: A modified device comfort scale using an 11-point rating overall score (0=Most Uncomfortable; 10=Most Comfortable).
Time Frame: Baseline
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1. NONE | Arm 2. BOOT | Arm 5. HFC | Arm 6. SAC
Number analyzed (Participants) | 17 | 17 | 17 | 17
score on a scale | 9.76 (0.44) | 7.82 (1.13) | 5.00 (2.62) | 5.12 (2.09)

5. Other Pre Specified Outcome: Participant Device Numerical Score
Description: A modified device comfort scale using an 11-point rating scale (0=worst assistive device;10=best assistive device).
Time Frame: over four sessions (an average of 2 hours for each session)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Arm 1. NONE | Arm 2. BOOT | Arm 5. HFC | Arm 6. SAC
Number analyzed (Participants) | 17 | 17 | 17 | 17
score on a scale | 9.06 (1.60) | 8.00 (1.37) | 6.35 (2.83) | 5.94 (1.95)

6. Other Pre Specified Outcome: Participant Device Preference
Description: The participant will rank in order (1-4) their preference of assistive device: NONE, BOOT, HFC and SAC.
Time Frame: one session (up to 2 hours long), out of 4 total sessions
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Arm 1. NONE | Arm 2. BOOT | Arm 5. HFC | Arm 6. SAC
Number analyzed (Participants) | 17 | 17 | 17 | 17
participants
  Preference 1 | 15 | 2 | 0 | 0
  Preference 2 | 0 | 13 | 3 | 1
  Preference 3 | 0 | 2 | 10 | 5
  Preference 4 | 2 | 0 | 4 | 11

ADVERSE EVENTS:
Time Frame: Each participant was assessed an average of one week.
Arm/Group | NONE, HFC+BOOT, SAC+BOOT, BOOT | NONE, BOOT, SAC+BOOT, HFC+BOOT | NONE, SAC+BOOT, BOOT, HFC+BOOT | NONE, BOOT, HFC+BOOT, SAC+BOOT | SAC+BOOT, NONE, BOOT, HFC+BOOT | SAC+BOOT, BOOT, NONE, HFC+BOOT | BOOT, NONE, SAC+BOOT, HFC+BOOT | BOOT, NONE, HFC+BOOT, SAC+BOOT | BOOT, HFC+BOOT, NONE, SAC+BOOT | HFC+BOOT, BOOT, NONE, SAC+BOOT | HFC+BOOT, NONE, BOOT, SAC+BOOT
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/2 | 0/2 | 0/1 | 0/3 | 0/1 | 0/2 | 0/2 | 0/2 | 0/2 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2 | 0/2 | 0/1 | 0/3 | 0/1 | 0/2 | 0/2 | 0/2 | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 0/2 | 0/2 | 0/2 | 0/1 | 0/3 | 0/1 | 0/2 | 0/2 | 0/2 | 0/2 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-11-23): https://cdn.clinicaltrials.gov/large-docs/63/NCT04978363/Prot_SAP_001.pdf